CLINICAL TRIAL: NCT05113992
Title: The Effect of Back Massage With Frankincense and Myrrh Oil Before the Cardiac Electrophysiological Procedure on Back Pain Intensity and Comfort
Brief Title: The Effect of Back Massage Before the Cardiac Electrophysiological Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, ülkü özdemir, assistant professor doctor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020/471
Record Dates: First submitted 2021-10-19; First posted 2021-11-09 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Massage
Keywords: Electrophysiological study; Comfort; Back Pain; Massage; Frankincense and Myrrh
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: 1. Intervention group 2. Placebo group 3. Control group. a randomized controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group massaged with frankincense and myrrh oil (Experimental): In the intervention group, 4% massage oil (3 ml jojoba fixed oil, 2% Frankincense and 2% Myrrh essential oil mixture) was applied on the skin on the forearm. Individuals who did not develop any reaction after thirty minutes and who met other inclusion criteria were included in the study. At the beginning of the study, the patient information form, VAS for back pain severity, and GCQ for comfort evaluation were applied by face-to-face interview method before the intervention. Then, in accordance with the massage application protocol, a back massage was applied for a total of 15 minutes, using 4% massage oil. Then EPS was applied to the individuals. VAS and GCQ were applied again at the 4th hour, which is the ambulation hour.
  Interventions: Other: aromatherapy massage
- . Placebo group massaged with jojoba oil, (Sham Comparator): In the placebo massage group, jojoba fixed oil was applied to the skin on the forearm. Individuals who did not develop any reaction after 30 minutes and who met other inclusion criteria were included in the study. At the beginning of the study, a patient information form, VAS for back pain severity, and GCQ for comfort evaluation were applied by face-to-face interview method before the intervention. Then, in accordance with the massage application protocol, a back massage was applied for a total of 15 minutes, using jojoba fixed oil. Then EPS was applied to the individuals. VAS and GCQ were applied again at the 4th hour, which is the ambulation hour.
  Interventions: Other: classic massage
- Control group (No Intervention): At the beginning of the study, a patient information form, VAS for back pain severity, and GCQ for comfort evaluation were applied by face-to-face interview method before the intervention. No intervention was applied to individuals in the control group. In order to ensure standardization between the groups, after 15 minutes of verbal communication, they were taken to the EPS process. After the procedure, VAS and GCQ were applied again at the 4th hour, which is the ambulation hour.

INTERVENTIONS:
Other: aromatherapy massage — In the intervention group, 4% massage oil (3 ml jojoba fixed oil, 2% Frankincense and 2% Myrrh essential oil mixture) was applied on the skin on the forearm
  Arms: Intervention group massaged with frankincense and myrrh oil
Other: classic massage — In the placebo massage group, jojoba fixed oil was applied to the skin on the forearm.
  Arms: . Placebo group massaged with jojoba oil,

SUMMARY:
This study was conducted to determine the effect of back massage with 4% frankincense and myrrh oil on back pain severity and comfort in patients who will undergo cardiac electrophysiological study (EPS).

DETAILED DESCRIPTION:
The study was conducted as a randomized controlled study. The population of the research consists of individuals who will undergo cardiac EPS in the angio unit of a heart hospital at a university. The sample size was determined as 20 people per group and a total of 60 people for an effect size of 0.131 and a power of 90%. Considering that there may be sample losses, 10 more patients were taken per group, and the study was completed with 30 patients for each group, a total of 90 people.

Randomization: Patients who met the inclusion criteria; They were assigned to one of three groups: 1. Intervention group massaged with frankincense and myrrh oil, 2. Placebo group massaged with jojoba oil, and 3. Control group. In hospital routine, patient appointments for the EPS procedure are determined on a weekly basis. Since the operation day of the research doctor who will perform the EPS procedure is Monday; Since patient rooms are not single occupancy; In addition, groups were randomized computer according to weeks to prevent contamination of frankincense and myrrh oil used for massage in the intervention group to the placebo and control groups.

Data were collected with the Patient Information Form, which includes the sociodemographic and health history of the individuals, the Visual Analogue Scale (VAS) for pain severity assessment, and the General comfort questionary (GCQ) for comfort.

Individuals who met the inclusion criteria in the study were assigned to the 1st Intervention group, 2nd Placebo group, and 3rd Control group in accordance with randomization, with their informed consent. No intervention was made in the standard treatment applied in the clinic.

In a systematic review and meta-analysis study, it is reported that bed rest is recommended for patients at wide intervals from 2 hours to 24 hours (2,4,6,12 and 24 hours) to prevent vascular complications after cardiac catheterization.Therefore, in this study, post-procedure back pain and comfort assessment were checked at the 4th hour, which is the clinical ambulation routine.

Interventions applied to the intervention group: In the intervention group, 4% massage oil (3 ml jojoba fixed oil, 2% Frankincense and 2% Myrrh essential oil mixture) was applied on the skin on the forearm. Individuals who did not develop any reaction after thirty minutes and who met other inclusion criteria were included in the study. At the beginning of the study, the patient information form, VAS for back pain severity, and GCQ for comfort evaluation were applied by face-to-face interview method before the intervention. Then, in accordance with the massage application protocol, a back massage was applied for a total of 15 minutes, using 4% massage oil. Then EPS was applied to the individuals. VAS and GCQ were applied again at the 4th hour, which is the ambulation hour.

Interventions Applied to the placebo group: In the placebo massage group, jojoba fixed oil was applied to the skin on the forearm. Individuals who did not develop any reaction after 30 minutes and who met other inclusion criteria were included in the study. At the beginning of the study, a patient information form, VAS for back pain severity, and GCQ for comfort evaluation were applied by face-to-face interview method before the intervention. Then, in accordance with the massage application protocol, a back massage was applied for a total of 15 minutes, using jojoba fixed oil. Then EPS was applied to the individuals. VAS and GCQ were applied again at the 4th hour, which is the ambulation hour.

Interventions Applied to the Control Group: At the beginning of the study, a patient information form, VAS for back pain severity, and GCQ for comfort evaluation were applied by face-to-face interview method before the intervention. No intervention was applied to individuals in the control group. In order to ensure standardization between the groups, after 15 minutes of verbal communication, they were taken to the EPS process. After the procedure, VAS and GCQ were applied again at the 4th hour, which is the ambulation hour.

Massage Application: Massage is the stimulation of soft tissues manually or mechanically. It is applied for therapeutic purposes such as maintaining blood and lymph circulation, relaxing muscles, reducing swelling, relieving pain, and providing sleep. The main maneuvers of classical massage are effleurage, petrissage, friction, tapotmen and vibration. In the study, effleurage, petrissage and friction were applied from these maneuvers. 15 to 45 minutes of massage therapy time. It has been reported to vary between. In this study, a 15-minute back massage was applied.

Massage application protocol: 1) The procedure is explained to the individual, his consent is obtained, 2) Hands are washed, gloves are worn, 3) The individual is given a comfortable sitting or lying position, 4) Curtain / screen is drawn or the room door is closed, 5) Back area for massage 6) 3 ml of massage oil is poured into the palms and fingers, 7) A total of 15 minutes of massage is applied by applying five minutes of effleurage, 5 minutes of petrissage, and 5 minutes of friction, 8) Gloves are removed, hands are washed and the process is recorded.

The data were evaluated in the statistical package program of IBM SPSS Statistics Standard Concurrent User V 26 (IBM Corp., Armonk, New York, USA). Descriptive statistics are given as number of units (n), percent (%), mean±standard deviation (x ̅±sd), median (M), first quartile (Q1) and third quartile (Q3). The normal distribution of the data of numerical variables was evaluated with the Shapiro Wilk test of normality and Q-Q graphs. Homogeneity of variances was evaluated with Levene's test. Comparisons between groups for the age variable were made with one-way analysis of variance, and between groups for procedure time and VAS values were made with Kruskal-Wallis analysis. The exact method of the chi-square test was used for the intergroup comparison of categorical variables. Comparison of scale scores between groups according to time was made with two-way analysis of variance in repeated measurements from general linear models. Bonferroni correction was applied to compare the main effects. A p value of <0.05 was accepted for statistical significance.

Ethics committee approval (decision no: 2020/471) from the Erciyes University Clinical Research Ethics Committee and written permission from the unit where the study would be conducted were obtained in order to conduct the study. In addition, those whose written consent was obtained through the Informed Consent Form were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are over 18 years old;
* agreeing to participate in the study;
* EPS planned from the femoral region;
* no communication problems (hearing, vision, speech, perception problems);
* According to VAS, there is no pain in any part of the body before the procedure;
* individuals who did not develop any reaction 30 minutes after applying the oils to be used on the skin on the forearm were included in the study.

Exclusion Criteria:

* Those who had an allergic skin reaction,
* skin disease in the back region,
* a history of fractures or surgical operations in the waist and back region in the last year,
* those who had neurological disorders (hemiparesis, etc.),
* those who received massage therapy in the last three months, those who were diagnosed with cancer,
* those who suffered from acute myocardial infarction were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | four hours
  It was used to evaluate the severity of back pain. The patient marks his or her own pain on a 10 cm ruler with painlessness (0) on one end and the most severe pain (10) on the other. The distance between the onset of "no pain" and this point marked by the patient is measured and recorded in centimeters. A high score indicates a high pain intensity.
General Comfort Questionary | four hours
  It was developed by Kolcaba in 1992. It was used to evaluate comfort. The scale is a four-point Likert type, positive and negative contains a total of 48 items. There are four sub-dimensions that physical, psychospiritual, environmental and sociocultural. The highest total score that can be obtained from the scale is 192, and the lowest total score is 48. The average value is determined by dividing the total score obtained by the number of scale items and the result is indicated in the 1-4 distribution. Low comfort is expressed by one and high comfort by four.

CONTACTS AND LOCATIONS:
Overall Officials: ülkü özdemir, Principal Investigator
Locations (1):
- Ülkü Özdemir, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
no planing